CLINICAL TRIAL: NCT03314532
Title: A Randomized Controlled Trial of the Efficacy of Hepatectomy or TILA-TACE in Patients With Resectable Hepatocellular Carcinoma
Brief Title: The Efficacy of Hepatectomy or TILA-TACE in Patients With Resectable Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAHZhejiangU-2017-071
Record Dates: First submitted 2017-10-08; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Surgical Resection; HCC
Keywords: Surgical Resection; TILA-TACE; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental design method will be adopted.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cases will be randomized by computer into the groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery group (No Intervention): We will completely resection of the visible tumor and made the resection margin negative. We will use regular/irregular resection of the liver tumor tissue, hemihepatectomy or extended hepatectomy.
- TILA-TACE group (Experimental): After femoral artery catheterization, 5-Fr angiography catheters will be used for complete radiography of the celiac artery, the hepatic artery proper, left and right hepatic arteries and their branches, and 2.8-Fr micro-catheters will be used for complete radiography of the tumor's nutrient arteries. Lipiodol-epirubicin emulsions and 5% sodium bicarbonate injection solutions will be used for perfusion of chemotherapy drugs. Different sizes of embolic microspheres will be used alternatively for chemoembolization.
  Interventions: Procedure: TILA-TACE

INTERVENTIONS:
Procedure: TILA-TACE — After femoral artery catheterization, 5-Fr angiography catheters will be used for complete radiography of the celiac artery, the hepatic artery proper, left and right hepatic arteries and their branches, and 2.8-Fr micro-catheters will be used for complete radiography of the tumor's nutrient arteries. Lipiodol-epirubicin emulsions and 5% sodium bicarbonate injection solutions will be used for perfusion of chemotherapy drugs. Different sizes of embolic microspheres will be used alternatively for chemoembolization.
  Arms: TILA-TACE group

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common cancers in the world with major occurrences in eastern Asian countries such as China. HCC is the third leading cause of cancer-related deaths in the world. There are multiple treatment options for liver cancer including surgery, transcatheter arterial chemoembolization (TACE), liver transplantation, absolute ethanol injection, radiation therapy, and biological therapy. Surgery is the primary radical treatment measure for HCC, but its indication is narrow and is only suitable for certain group of patients. Another common treatment for liver cancer, TACE, can not only block tumor blood supply, control tumor growth, or even cause necrosis and result in tumor shrinkage, it can also deliver target chemotherapy drugs to the tumor tissue. However, there are still some controversies on the efficacy of TACE treatment. Therefore in this study, we will conduct a randomized comparison study of the efficacy of surgical resection and TILA-TACE treatment.

DETAILED DESCRIPTION:
The Barcelona Clinic Liver Cancer staging system (BCLC) is one of the more recognized staging criteria and has been recommended by the European Association for the Study of Liver and the American Association for the Study of Liver Diseases. BCLC staging is based on patients' general condition, tumor condition, and liver function to identify the best treatment option and predict prognosis using evidence-based medicine. Surgical excision is recommended for BCLC stage 0, liver transplantation or radiofrequency ablation is recommended for BCLC stage A, and TACE treatment is recommended for BCLC stage B.

However, there are still some controversies on the efficacy of TACE treatment. In recent years, development of technologies has led to improved methods including targeting-intratumoral-lactic-acidosis TACE (TILA-TACE). Early clinical practice has confirmed that compared with TACE, TILA-TACE has a relatively high response rate and efficiency. In clinical practice, the current standard treatments for patients with surgically resectable HCC are controversial and there is no recommendation in the guidelines.

This study is designed to evaluate and compare the therapeutic efficacies of surgical resection and TILA-TACE treatment in patients with resectable HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75 with no gender, ethnicity, religion, or geographical restrictions.
2. Diagnosed HCC patient.
3. The following criteria will be used for the evaluation of tumor resectability and adequate remaining liver volume: ≥ 30% remaining liver volume/total liver volume for non-hepatitis patients; ≥ 40% remaining liver volume/total liver volume for hepatitis patients.
4. Imaging examination with no cancer embolus above the secondary branch of the portal vein.
5. New lesions found five years after liver cancer treatment.
6. Child-Pugh A or B grade liver function.
7. No concurrent malignancies in other systems.
8. Informed subjects who fully understand and willingly cooperate with the test program with signed relevant documents.

Exclusion Criteria:

1. Suffer from other malignancies.
2. Have received any other liver cancer treatments.
3. Pathological diagnosis as non-HCC.
4. Experience large blood vessel invasion, distant metastases, or unresectable liver cancer.
5. One or more organ failures.
6. Child-Pugh C grade liver function.
7. Incomplete surgical resection or TILA-TACE.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
disease-progression-free period | This will be the time period from the beginning of treatment to the time that disease progression has been observed (up to 120 months).
  This will be the time period from the beginning of treatment to the time that disease progression has been observed.

SECONDARY OUTCOMES:
overall survival period | from the beginning of the treatment, until the death of the patient or the end of the study period (up to 100 months).
  from the beginning of the treatment, the follow-up, until the death of the patient or the end of the study period, as well as the 1-year, 3-year, and 5-year survival rates.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang-tao Li, MD, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sastre J, Diaz-Beveridge R, Garcia-Foncillas J, Guardeno R, Lopez C, Pazo R, Rodriguez-Salas N, Salgado M, Salud A, Feliu J. Clinical guideline SEOM: hepatocellular carcinoma. Clin Transl Oncol. 2015 Dec;17(12):988-95. doi: 10.1007/s12094-015-1451-3. Epub 2015 Nov 25. PMID 26607931
- [Result] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Result] Chao M, Wu H, Jin K, Li B, Wu J, Zhang G, Yang G, Hu X. A nonrandomized cohort and a randomized study of local control of large hepatocarcinoma by targeting intratumoral lactic acidosis. Elife. 2016 Aug 2;5:e15691. doi: 10.7554/eLife.15691. PMID 27481188
- [Result] Zhou WP, Lai EC, Li AJ, Fu SY, Zhou JP, Pan ZY, Lau WY, Wu MC. A prospective, randomized, controlled trial of preoperative transarterial chemoembolization for resectable large hepatocellular carcinoma. Ann Surg. 2009 Feb;249(2):195-202. doi: 10.1097/SLA.0b013e3181961c16. PMID 19212170